CLINICAL TRIAL: NCT02272075
Title: Image Comparison of a Mobile Colposcope (SmartScope) vs. a Standard Colposcope for Directing Cervical Biopsies in Women With Abnormal Pap Smears: A Non-inferiority Trial.
Brief Title: SmartScope vs Standard Colposcope for the Evaluation of Cervical Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Bruce Kahn, MD, Scripps Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Scripps-Mobile OCT 1
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer
Keywords: screeening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- active colposcope (Active Comparator): Mobile OCT M3 scope
  Interventions: Device: Mobile OCT M3 scope
- Standard of Care (No Intervention): Standard of Care

INTERVENTIONS:
Device: Mobile OCT M3 scope
  Arms: active colposcope

SUMMARY:
This trial will compare images obtained from a mobile colposcope with those obtained using a standard of care.

DETAILED DESCRIPTION:
This trial will compare images obtained from a mobile colposcope with those obtained using a standard colposcope in women with abnormal pap smears. It is a non-inferiority trial. Blinded images will be evaluated be experts in colpsocopy and compared

ELIGIBILITY:
Inclusion Criteria: abnormal cervical cancer screening by pap smear of high risk HPV test -

Exclusion Criteria: no consent

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
image non-inferiority | 6 months
  imafge non-inferiority

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kahn, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic, San Diego, California, United States